CLINICAL TRIAL: NCT05183685
Title: Outcomes of a Risk Assessment and Management Program Using Telecare Consultation Among Patients With Diabetes Mellitus in General Out-patient Clinic: A Hybrid Effectiveness-implementation Study
Brief Title: a Risk Assessment and Management Program Using Telecare Consultation Among Patients With Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Arkers, Wong, Assistant professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: A0034230
Record Dates: First submitted 2021-12-07; First posted 2022-01-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; telecare consultation
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants will receive alternative telecare consultation and face to face consultation every 14 weeks.
  Interventions: Procedure: telecare consultation
- Control group (Placebo Comparator): The participants will receive usual face to face consultation every 14 weeks.
  Interventions: Procedure: Usual face to face consultation

INTERVENTIONS:
Procedure: telecare consultation — Participants will use zoom to communicate with the doctors in clinic.
  Arms: Intervention group
Procedure: Usual face to face consultation — Participants will have face-to-face communication with the doctors in clinic.
  Arms: Control group

SUMMARY:
Telecare consultation, which is defined as a two-way synchronized visual (voice and image) communication between patients and healthcare professionals using telecommunication applications such as Zoom, has become a major trend in recent years. The current COVID-19 pandemic provides an impetus to drive change and increase the uptake of telecare consultation in healthcare. To the best of investigators' knowledge, there is no translational research available that simultaneously implements and evaluates the telecare model of care delivered in a primary care setting. The present study will be the first in Hong Kong to fill this service and knowledge gap in the care of DM patients.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or above, having a confirmed diagnosis of diabetes, having regular follow-ups in the clinic

Exclusion Criteria:

* having dementia, having unaccompanied hearing or vision loss, not having an Internet connection at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 780 (Actual)
Dates: Start 2022-12-10 (Actual); Primary Completion 2025-08-31 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
HbA1c, defined as the amount of blood sugar attached to hemoglobin. | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  An HbA1c test shows what the average amount of glucose attached to hemoglobin has been over the past three months. It's a three-month average because that's typically how long a red blood cell lives. The blood glucose level will be measured at baseline pre-intervention, 42 weeks, and 84 weeks by a doctor.

SECONDARY OUTCOMES:
Fasting lipid profile that will be drawn by patient's blood. The profile includes high and low-density lipoprotein, cholesterol level, and triglyceride level | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  Investigators are measuring the change of high- and low-density lipoprotein, cholesterol level, triglyceride level
body mass index, defined as the weight in kilograms divided by height in meters. | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  the change of weight in kilograms divided by height in meters
Medication adherence | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  the change of Medication adherence will be determined using the Adherence to Refills and Medications Scale. This 12-item scale has a total score ranged from 12 to 48, with lower scores representing better medication adherence.
Quality of life, defined by the standard of health, comfort, experienced by diabetic patients, which is measured by SF-12 questionnaire. SF-12 questionnaire can measure the physical and mental health components of quality of life among diabetic patients. | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  Investigators will measure the change of physical and mental health components of quality of life of participants, measured by the Chinese version of Short-form 12-item version 2 scale.The 12 items in the questionnaire included two from each of the physical functioning (PF), role limitation due to physical problems (RP), role limitation due to emotional problems (RE), and mental health (MH) scale and one item from each of the bodily pain (BP), general health (GH), vitality (VT), and social functioning (SF) scale of the original SF-36 questionnaires. The items in the questionnaire were rated on Likert-type scales and summed to provide easily interpretable scales for physical and mental health components. Higher scores indicated better quality of life.
Number of attendances at a general practitioners' office, emergency department, hospital, and general out-patient clinic | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  To measure the utilization of healthcare services by stroke patient before and after the intervention.

OTHER OUTCOMES:
Reach, which means reach into the target population. It measures the number of patients who are eligible to receive telecare consultation, excluded, invited. | 84 weeks (T3)
  the number of patients who are eligible to receive telecare consultation, excluded, invited to participate, and enrolled in the study
Adoption, which means adoption by the staff and setting. It measures the user readiness for the program adoption | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  Use Readiness for Implementation Model Survey to evaluate the adoption success of telecare consultation.
Implementation. It measures the fidelity of the program | baseline pre-intervention (T1), 42 weeks (T2) and 84 weeks (T3)
  Use performance checklist to evaluate whether each task of the intervention has been implemented according to the protocol
Maintenance. It measures the sustained effect of the program. Cost-effectiveness will be measured by calculating the cost used in both groups. | 84 weeks (T3)
  Cost evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Tuen Mun Hospital, Tuenmen, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong AKC, Liu LZ, Wong FKY, Liang J, Tong DWK, Chan ML, Wong MK, Wong BC, Tang CYS, Ho WH, Chiang SC. Voices from the field: healthcare professionals' insights on sustaining telemedicine for diabetes management in Hong Kong primary care. Front Digit Health. 2025 Nov 28;7:1665424. doi: 10.3389/fdgth.2025.1665424. eCollection 2025. PMID 41395628